CLINICAL TRIAL: NCT00371839
Title: Clinical Applications for Time-Compressed Speech Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4338-R
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2014-11-19 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Hearing Loss
Keywords: Hearing Loss; Hearing Aids; Rehabilitation of hearing impaired
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild Hearing Loss (Active Comparator): Audiological Evaluation will show average hearing threshold at 500, 1000, 2000, and 4000 Hz of 20-39 decibels hearing level (dBHL)
  Interventions: Procedure: Audiological Evaluation
- Moderate Hearing Loss (Active Comparator): Audiological Evaluation will show average hearing threshold at 500, 1000, 2000, and 4000 Hz of 40-49 decibels hearing level (dBHL)
  Interventions: Procedure: Audiological Evaluation
- Moderate-Severe Hearing Loss (Active Comparator): Audiological Evaluation will show average hearing threshold at 500, 1000, 2000, and 4000 Hz greater than 50 decibels hearing level (dBHL)
  Interventions: Procedure: Audiological Evaluation

INTERVENTIONS:
Procedure: Audiological Evaluation — Tests of hearing, cognition, and speech perception

SUMMARY:
The purpose of this study is to determine the effects of age-related cognitive changes on hearing aid benefit based on hearing aid compression time constants.

The hypothesis is that people with poor working memory skills will benefit from slow time constants in hearing aid compression while those with good working memory skills will be able to benefit from more sophisticated compression algorithms with rapid time constants.

DETAILED DESCRIPTION:
Recent research has shown the relevance of cognitive function in hearing aid evaluation and the sensitivity of the aging auditory system to temporal distortions. The proposed investigation will examine the interaction of working memory and hearing aid compression method on speech recognition in background competition for older listeners. This interaction will be investigated for the following three forms of background competition:

1. Competition from continuous speech-shaped noise.
2. Competition from speech-modulated noise.
3. Competition from a single interfering talker.

The goals of the study will be accomplished in two phases. In the first phase, 160 adults aged 50 through 75 years will be evaluated on a battery of tests to determine their cognitive capacity, time-compressed speech scores and their candidacy for inclusion in the second phase of the study. At the conclusion of this phase of testing, the participants will be divided into three groups:

1. subjects with TCS test scores in the highest quartile (the HIGH group)
2. subjects with TCS test scores in the lowest quartile (the LOW group)
3. the remaining listeners

The second phase of the experiment will include listeners from the HIGH and LOW groups only. These subjects will be evaluated with respect to their speech recognition ability for three types of interference (steady-state noise, speech-modulated noise, single interfering talker). The HINT test (Nilsson, Soli, & Sumida, 1995; Nilsson et al., 1994) will be used to obtain the signal-to-noise ratio (SNR) at 50% recognition for the three masking conditions for each of three types of amplification:

1. one- channel linear amplification (LINEAR) with frequency shaping
2. two-channel wide dynamic range compression with fast time constants (FAST)
3. two-channel wide dynamic range compression with slow time constants (SLOW) Listener groups will be compared across hearing aid conditions and across background interference conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 50 to 75 years old.
* Hearing loss will be limited to 40 dB HL from 250 Hz through 1000 Hz, and to 60 dB HL through 4000 Hz.
* Hearing loss must be greater than 25 dB at two or more frequencies from 250 to 4000 Hz.

Exclusion Criteria:

* None of the participants will be current or past hearing aid users; all will be free of ear disease.
* Participants with conductive hearing losses, defined as air-bone gap greater than 15 dB, will be excluded.
* The audiometric battery with acoustic reflex thresholds and decay measurements will be used to exclude anyone with evidence of a central disorder or a pathology other than a sensorineural loss. Those potential participants will be referred to a medical professional.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie R. Leek, PhD, Principal Investigator — VA Loma Linda Healthcare System, Loma Linda, CA

REFERENCES:
- See also: This is the web page of the VA research Center where the study took place — http://www.ncrar.research.va.gov/Index.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans from 50 to 75 years of age with hearing loss, not hearing aid wearers
Pre-assignment Details: After audiometric thresholds were tested, subjects were assigned to one of three groups based on their pure tone averages (PTA) of thresholds at 500, 1000, 2000, and 4000 Hz. The groups were:
  Mild (PTAs of 20-39 decibels (dB) hearing level (HL) Moderate (PTAs of 40-49 dB HL) Moderate-Severe (PTAs over 50 dB HL)
Groups:
- Mild HL: Average hearing loss between 20 and 39 decibels hearing level (HL)
  Study performance on cognitive and hearing tests
  Audiological Evaluation: Tests of hearing, cognition, and speech perception
- Mod HL: Average hearing loss between 40 and 49 decibels hearing level (HL)
  Study performance on cognitive and hearing tests
  Audiological Evaluation: Tests of hearing, cognition, and speech perception
- ModSev HL: Average hearing loss greater than 50 decibels hearing level (HL)
  Study performance on cognitive and hearing tests
  Audiological Evaluation: Tests of hearing, cognition, and speech perception
Period: Overall Study
Arm/Group | Mild HL | Mod HL | ModSev HL
Started | 49 | 20 | 9
Completed | 32 | 13 | 7
Not Completed | 17 | 7 | 2
Not completed — Death | 4 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 4 | 0
Not completed — Lost to Follow-up | 6 | 3 | 2

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Mild HL | Mod HL | ModSev HL | Total
Number analyzed (Participants) | 32 | 13 | 7 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (6.8) | 62.7 (7.0) | 65.1 (5.1) | 61.7 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 31 | 12 | 6 | 49

OUTCOME MEASURES:

1. Primary Outcome: Ability to Understand Speech in Noise Background
Description: Measure speech perception for sentences in background noise
Time Frame: one year
Measure: Mean (Standard Deviation); unit: Percent correct of 100 presented words
Arm/Group | Mild HL | Mod HL | ModSev HL
Number analyzed (Participants) | 32 | 13 | 7
Percent correct of 100 presented words | 84 (4.0) | 78 (7.0) | 47 (9.0)

ADVERSE EVENTS:
Description: 9 subjects were lost to followup and could not be contacted for continued data collection
Groups:
- Arm 1: Study performance on cognitive and hearing tests
  Audiological Evaluation: Tests of hearing, cognition, and speech perception
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 6/69
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=69)
Death or terminal illness (General disorders) | 6 — Upon attempting to schedule an experimental session, the study team was notified of death or terminal illness of a participant, not related to study participation. No cause of death or type of illness were reported to the team.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes